CLINICAL TRIAL: NCT05232721
Title: Evaluation of a Point-of-care Testing Instrument for Fecal Immunochemical Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Clinical Professor, Shandong University
Other Study IDs: 2022SDU-QILU-105
Record Dates: First submitted 2022-01-06; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fecal Immunochemical Test: People in this group will detect hemoglobin in stool before colonoscopy by the new instrument
  Interventions: Diagnostic Test: The new instrument and colonoscopy with pathological examination

INTERVENTIONS:
Diagnostic Test: The new instrument and colonoscopy with pathological examination — Detect hemoglobin in stool by the point-of-care testing instrument before colonoscopy, detect colon lesion using colonoscopy and pathological examination.

SUMMARY:
Early detecting and removing of colorectal advanced adenomas can reduce incidence of colorectal cancer.Use of the fecal immunochemical test (FIT) for colorectal cancer (CRC) prevention is supported by previous studies.However existing instruments have low portability.The purpose of this study is to test the performance of a Point-of-care testing instrument for fecal Immunochemical test(FIT) .

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer worldwide and has become a progressively important public health problem that inevitably leads to an increase in morbidity and medical costs. Therefore, many countries have a screening program in place to lower the incidence of CRC. Subjects with a positive fecal immunochemical test (FIT) have a much higher likelihood of advanced neoplasms than the general population.However existing instruments have low portability.The purpose of this study is to test the performance of a Point-of-care testing instrument for fecal immunochemical test (FIT).

ELIGIBILITY:
Inclusion Criteria:

* People who use the new instrument for fecal immunochemical test(FIT)
* People sign an "informed consent form"

Exclusion Criteria:

* People with history of surgery in any part of the large bowel;
* People with symptoms including visible rectal bleeding, hematuria, hemorrhoid bleeds, severe and acute diarrhea and 7th type stool (Bristol feces score);

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People who use the new instrument for Fecal Immunochemical Test.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of advanced neoplasms | 4 months
  The study is committed to test the diagnostic efficacy of the new instrument to advanced neoplasms.We will measure the sensitivity and specificity of the instrument

SECONDARY OUTCOMES:
Diagnostic performance of Colorectal Cancer | 4 months
  The study is committed to test the diagnostic efficacy of the new instrument to colorectal cancer.We will measure the sensitivity and specificity of the instrument

CONTACTS AND LOCATIONS:
Overall Officials: Li yanqing, Professor, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China